CLINICAL TRIAL: NCT06449261
Title: C5-C6 and Thoracic Spine Mobilization With Postural Correction Exercise Compared With Conventional Therapy in Patients With Adhesive Capsulitis - A Two-group, Parallel-arm, Single-blinded, Randomized Clinical Trial
Brief Title: Manual Therapy of Spine With Postural Correction Exercise Compared With Conventional Therapy in Patients With Adhesive Capsulitis - A Randomised Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-FAC-134-MAY-2024
Record Dates: First submitted 2024-05-11; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-03

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: A two-group, parallel-arm, single-blinded, randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receives C5-C6 and thoracic spine mobilization with postural correction (Experimental): The patient will be made to lie in a prone position with the therapist beside her/his height- adjusted couch. Then the therapist who is certified to provide manual therapy will impart grade III+ posterior-to-anterior mobilization/lateral glide according to Maitland class cation focused on the cervical spine, C5-6 segment for 3 bouts of 30 seconds/2 days in a week for 3 weeks. Followed by the patient will be permitted to rest for a few minutes less than 10 minutes before starting the thoracic mobilisation. Thoracic mobilisation will be administered both at central and unilateral postero-anterior passive accessory intervertebral motions (PAIVMs) based on manual therapy evaluation at the thoracic spine.
  Interventions: Other: Spinal Manual therapy used in Physiotherapy Practice
- Group receives conventional therapy (Active Comparator): Controls will receive ultrasound therapy, passive shoulder mobilisation focussed at Glenohumeral joint, self-stretching exercises and patient education by qualified therapist according to clinical practice guidelines while the experimental group underwent spine mobilization with postural correction exercises for 3 weeks.
  Interventions: Other: Spinal Manual therapy used in Physiotherapy Practice

INTERVENTIONS:
Other: Spinal Manual therapy used in Physiotherapy Practice — C5-C6 and thoracic spine mobilization with postural correction

SUMMARY:
Adhesive capsulitis (AC) is often self-limited but can persist for years and may never fully resolve. The most effective treatment for adhesive capsulitis is uncertain till date. Though neural links are being studied on one side and postural alteration too was postulated to cause shoulder pathology. However, the effectiveness of C5-C6 and thoracic spine mobilization with postural correction remains unexplored in the treatment of AC. This study aimed to investigate whether C5-C6 and thoracic spine mobilization with postural correction are more effective than conventional therapy in pain, range of motion(ROM), and disability in patients with AC. The outcome of the study must provide valid information to enhance the prognostic value of adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis (AC) is often self-limited but can persist for years and may never fully resolve. The most effective treatment for adhesive capsulitis is uncertain till date. Though neurological control of the shoulder girdle muscles is mainly from cervical roots, particularly from C5/C6 roots, there was not sufficient research to associate this link with AC. Evidence confirms that there is an association between posture and shoulder mobility. However, the effectiveness of C5-C6 and thoracic spine mobilization with postural correction remains unexplored in the treatment of AC. We aimed to investigate whether C5-C6 and thoracic spine mobilization with postural correction are more effective than conventional therapy in pain, range of motion(ROM), and disability in patients with AC.

Methods The protocol is written according to the SPIRIT statement to enhance transparency of content and completeness. Two-group, randomized controlled trial with blinded assessors. A total of 66 adults with AC will be randomly assigned to experimental group to receive C5-C6 and thoracic spine mobilization with postural correction sessions (n=33) and the others(n=33) in control group to receive conventional therapy within a period of 3 weeks. Primary outcomes are Shoulder Pain, range of motion (ROM) of the shoulder joint and Disability Index (SPADI) were to be measured at pre, postintervention following 3 weeks and 3 months..

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AC & a Positive for Apley's scratch test.
* Adhesive capsulitis (with symptoms for at least three months and less than 12 months[18]
* Both Gender
* Age 27-70
* Sleep-disturbing night pain

Exclusion Criteria:

* Patients who are unwilling to participate
* patients with malignancy
* AC Secondary to fracture and uncontrolled hypertension.
* Unstable cardiac conditions
* Patient with neurological conditions
* Patient with reported concurrent cervical issues

Ages: 27 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Range of motion of shoulder | 1 Year
  The smartphone clinometer (Plaincode Software Solutions) is readily available at low cost for several smartphones, including the iPhone, which will be used by all examiners in this study
SPADY scale | 1 Year
  In the original version, the patient was instructed to place a mark on the VAS for each item that best represented their experience of their shoulder problem over the last week [26]. Each subscale is summed and transformed to a score out of 100. A mean is taken of the two subscales to give a total score out of 100, a higher score indicating greater impairment or disability.
Cervical Range of motion | 1 Year
  Clinometer app on smartphones is a reliable and valid device for assessing cervical flexion, extension, lateral flexion, and rotation. The results from the study demonstrated moderate to excellent (ICC = .87-.96) concurrent validity in all 6 cervical movements when compared with the universal goniometric measurements

CONTACTS AND LOCATIONS:
Overall Officials: Watson Arulsingh D R, PhD, Principal Investigator — Gulf Medical University
Locations (2):
- United Arab Emirates (2):
  - Sharad, Al Jurf, Ajman Emirate
  - Thumbay Hospital, Ajman

IPD SHARING:
Plan to Share IPD: No